CLINICAL TRIAL: NCT04583670
Title: How Point-of-care Ultrasound Affects the Diagnostic and Therapeutic Process in General Practice. A Prospective Follow-up Study in France
Brief Title: Point of Care Ultrasound Use by General Practitioners in France (Echo-MG)
Acronym: Echo-MG
Status: Completed | Type: Observational
Sponsor: Sorbonne University (Other)
Collaborators: Aalborg University (Other); Agence Regionale de Sante d'Ile de France (Other Government)
Responsible Party: Principal Investigator, Gladys IBANEZ, Head of General Medicine Department, Sorbonne University
Other Study IDs: Echo-MG
Record Dates: First submitted 2020-10-05; First posted 2020-10-12 (Actual); Results first posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Point of Care Ultrasound
Keywords: ultrasound; primary care; diagnostic; general practice; physical examination; family medicine
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient physical examination with ultrasound: No intervention

SUMMARY:
This study explores how Point of Care Ultrasound (POC-US) is used in general practice in France and how it affects the diagnostic process and treatment of patients.

General practitioners (GPs) will register information each time they use POC-US during a one month period.

The aim of this study is to describe the use of POCUS and its role in the diagnostic and therapeutic process in general medicine.

* Description of the use of POCUS through indication, organs scanned, findings, frequency , time consumption.
* Analysis of the role of POCUS in the diagnostic process: change of diagnostic hypotheses and change of certainty in the main diagnostic hypothesis.
* Analysis of the role of POCUS in the therapeutic process: change in the care pathway and the therapeutic initial plan.

This is an observational study without any intervention.

DETAILED DESCRIPTION:
There are few studies describing the use of POCUS in general medicine. Most of them are descriptive studies made more than ten years ago while recent technological development has resulted in better quality images. There is no study with high level of evidence, and the majority of the literature is made of descriptive reports based on the activity of a small number of physicians.

Unlike other countries, France has currently no recommendations on the modalities of use for POCUS. There are no guidelines on the GP curriculum nor on the appropriate equipment for general practitioners, nor on the certification process.

In the current state of knowledge, it seems relevant to establish an overview of the practice of POCUS in general medicine in France. This work is part of an international European reflection on the use of POCUS in general practice and its role in the diagnostic process, therapeutic process and the patients' care pathway in Denmark, in Norway and in France.

The current protocol was written in collaboration with the GP Research Unit of Aalborg. The Danish protocol was completed between January 2018 and July 2019 in Denmark, registered at clinicaltrials.gov NCT03375333. This part of the protocol constitutes the French study.

The aim of this study is to describe the use of POCUS and its role in the diagnostic and therapeutic process in general medicine.

Description of the use of POCUS through indication, organs scanned, findings, frequency, time consumption.

Analysis of the role of POCUS in the diagnostic process: change of diagnostic hypotheses and change of certainty in the main diagnostic hypothesis.

Analysis of the role of POCUS in the therapeutic process: change in the care pathway and the therapeutic initial plan.

The study is a prospective observational cohort study. It will take place in France among 30 GPs that use POCUS during consults in their office or during home visits.

Any patient having a POCUS scan during a consultation by a participant GP may be included in the study. Patients will be informed and asked to sign a consent form before inclusion in the study. Patients will be informed of the study terms by their GP and through an information note in the waiting room. Patients will be excluded if they refuse to participate in the study or are unable to give informed consent. Refusal to participate in the study will not change patient management.

There will be no intervention in this study. The GPs already use ultrasound during their physical examination. The data recorded for this study will reflect the daily practice of general practitioners using POCUS. There will be no additional exams or other ways to change the patient management. If a second POCUS is performed later for the same patient, this data will not be collected. Only data from the patient's first examination will be collected.

Each investigator will collect data about every POCUS examination performed during the inclusion period of 22 consecutive working days.

The data collection tool is based on the questionnaire originally developed by the Center for General Practice at Aalborg University in Denmark from literature data, a dialogue with the "Ultrasound group of the Danish College of General Medicine" and an interview study. The registration tool was developed as a questionnaire to be used before and after the GP uses POCUS in the consultation. A time log is included to ensure that the questionnaire has been completed before and after the exam.

For this study, the questionnaire will first be translated into French and then back-translated (reverse French-English translation) by two bilingual translators separately. The result of the back-translation will be analyzed and a second French version will be submitted to French general practitioners practicing POCUS and members of the "Ultrasounds group of the College of General Medicine" in France. For each theme of the questionnaire, there will be a common part of questions, to ensure the comparability of the results between the different European countries. An additional set of questions relevant to general practice in France will be discussed and validated by the French College of General Medicine. The acceptability and validity of the questionnaire will be tested during focus groups and a pilot study.

The GPs will be asked to fill a questionnaire in the online database SurveyXact each time they use POCUS during their daily work. The data will be registered electronically in SurveyXact with a time log to ensure a before and after registration.

The GPs can access the questionnaire on their mobile phone, iPad or computer, using a unique link (respondent link) allocated to each participant. A key file, connecting each GP participant with the respondent link in SurveyXact (link), will be safely stored at Center for General Practice at Aalborg University, Denmark.

The GPs will give each patient a unique ID-number. A key file connecting this ID-number and the patient's identity will be safely stored at the GP's clinic.

There will be a registration of the date and time, when the GP starts filling the questionnaire and finishes the final question. Furthermore, a variable with the exact time between "before" and "after" questions will be created. If GPs use less than one minute on this page and the GP registers a duration of the POC-US > 1 minute, there will be no "before and after" registration, but only an "after" registration. In that case, the "before" answers will be excluded.

Participants retention In order to calculate the participant retention rate, defined by the proportion of eligible patients included in the study, GPs will be asked to record age and gender for each patient eligible but not included in the study (time constraints, patient refusal or other reasons).

Data management Data will be saved electronically on the SurveyXact server and on a server at Aalborg University and will only be accessed by the research group using personal passwords. The patient key file and consent forms will be safely stored at the GPs' office and the research group will not have access to this information during the study.

Any paper editions of the registration tool or questionnaire (in case of server breakdown) will be safely stored at the GPs office until the end of the data collection. Afterwards, they will be safely stored at the General Practice Department of Sorbonne University, 27 rue de Chaligny, PARIS 75012, FRANCE.

The use of ultrasound will be described in terms of ultrasound indications, organs explored, findings, frequency of use and duration of the examination.

The indications of POCUS will be described through the GP's intention regarding ultrasound:

* to answer a specific clinical question (yes / no / maybe) and document the answer in the medical file
* to conduct therapeutic education
* to monitor or control an ultrasound finding
* to screen an asymptomatic patient
* to scan to improve technical ultrasound skills without any clinical profit
* to perform a diagnostic scan with a detailed description of anatomical regions and provide a complete diagnostic report.

The frequency of the different POCUS examinations will be summarized in relation to the organs scanned. The performed POCUS examinations are defined as organs scanned and not as standardized procedures such as FAST, FATE or LUS since there might be differences in the definition and interpretation of these examinations. The organs scanned are registered on a list of organs in the questionnaire. The possibilities in this list originate from interviews with GPs using POCUS and from Danish pilot testing. This list will be discussed during a focus group of French GPs using POCUS. The GPs will be allowed to write in free text if organs are missing from the list.

The frequency of POCUS use will be described as the number of GP consultations where POCUS is used over the total number of GP consultations per day during 22 consecutive working days.

Each participant will provide information on the total number of face-to-face consultations she or he has had during the study period. If the GP uses a portable or ultraportable ultrasound device during home visits, they will be included in the total number of consultations.

The GPs will measure the time used for the POCUS examination. The time registration starts when the scanning begins and ends when the scanning has been finished. Hence, it will only include the duration of the POC-US examination, not information about the scanning or other elements of the consultation. This time registration will be described in minutes for each type of POC-US examination.

The study will describe the main diagnostic hypothesis recorded before and after POCUS, the total number of diagnostic hypotheses recorded before and after POCUS, the change in the total number of diagnoses hypotheses, the change in the GP's confidence in the diagnostic hypotheses (5-point Likert scale). To test the reliability of the GP confidence in the diagnoses, we will describe the correlation between the GP's confidence and the type of organ scanned, the change from a symptom diagnosis to a disease diagnosis and the decrease in the number of diagnostic hypotheses. A scatter plot will be used to describe the relationship between "confidence in the main diagnostic hypothesis" and "the number of diagnostic hypotheses". Frequency of incidental findings will be described separately related to the organs explored.

After the use of POCUS, the GPs will be shown their "Before-POCUS" diagnostic hypothesis and asked if these diagnoses have changed. If the diagnoses have changed, they will be asked to specify them.

The diagnostic hypotheses are registered as detailed free text in the questionnaire. The corresponding ICPC-2 (International Classification of Primary Care-2) codes will be coded from the free text by the research team.

The observed change in the diagnostic hypotheses will be described by the frequency of declared diagnostic hypotheses changes and the overall registered change in the ICPC-2 codes.

The patient's plan before and after POCUS and the planned treatment before and after POCUS will be described. The analysis will describe the relationship between the ultrasound findings and the change in the patient management (diagnostic process, treatment, care pathway). The diagnostic and therapeutic modifications will be described by the frequency of responses or by the change in the total number of responses.

The statistical analysis will be descriptive. Data collection will mainly be done using nominal variables. However, the variable "GP's confidence in the diagnostic hypotheses" will be measured by an ordinal variable, "the duration of the examination" and "the patient's age" by a continuous variable.

If the continuous variables follow the normal distribution, they will be described with means and either a standard deviation or a 95% confidence interval of the mean. If they are not normally distributed, they will be described with a median and interquartile range.

To assess the relationship between paired variables the Mac Nemar test will be used. To compare the characteristics of included and excluded patients, a Chi-2 test will be used. Results will be considered statistically significant if the p-value is less than 0.05. For highly significant results with p-values much lower than 0.05, we will simply report p < 0.01.

After using POC-US the GP is shown the "before POC-US plan for the patient" and asked if this plan has changed. If the plan has changed, the GP is asked to specify.

Change in the plan for the patient is defined as the frequency of declared change after registration from one possible answer to another or change in the total number of possible answers.

After using POCUS, the GP is shown the "before POC-US planned treatment for the patient" and asked if this planned treatment has changed. If the planned treatment has changed, the GP is asked to specify.

Change in the planned treatment of patients is defined as the frequency of declared change described before and after registration from one possible answer to another, or in the total number of possible answers.

ELIGIBILITY:
Inclusion Criteria:

* minimum use of POCUS on two anatomical areas
* GP activity for minimum two days / week
* A minimum of two scanning probes
* Previous participation in formal education in the use of POC-US
* Minimum six-month experience with POCUS in general practice.
* Estimated use of POCUS on a daily basis (average)

Exclusion Criteria:

* Conflict of interest, e.g. if the GP is part of the research group or if the GP has/had direct financial interest in selling ultrasound devices.
* If less than five patients have been enrolled

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: General practitioners practicing POCUS in rural or urban areas, alone or in groups with fixed or portable devices will be eligible.
Sampling Method: Non-Probability Sample
Enrollment: 655 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mariela Skendi, MD, MSc, Study Director — General Practice Department Sorbonne University; Roxane Liard, Principal Investigator — General Practice Department Sorbonne University
Locations (17):
- France (17):
  - Cabinet de médecine générale, Le Pecq, France
  - Centre Erdian SOS Médecins, Anglet
  - Maison de santé, Avon
  - Cabinet médical, Conches-en-Ouche
  - Maison Médicale, Égly
  - CMS Salvador Allende, La Courneuve
  - Cabinet médical, Limay
  - Cabinet médical, Mirabeau
  - Cabinet IPSO, Paris
  - Cabinet médical, Paris
  - Maison médicale, Pont-Croix
  - Cabinet médical, Saint-Etienne
  - Cabinet médical, Saint-Médard-en-Jalles
  - Maison médicale, Saint-Nom-la-Bretêche
  - Cabinet médical, Strasbourg
  - Cabinet médical Le Vallet, Vallet
  - SOS médecins, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: Yes
The data registered are available for the cooperating researchers at the university in Aalborg Denmark. The purpose of further analyses is to compare the external validity of the questionnaire.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2025
Access Criteria: The data are only available for collaborating researchers at the Center for General Practice, University of Aalborg, Denmark. The principal investigator will have access to pseudo-anonymized data registered on the online platform.

REFERENCES:
- [Background] Moore CL, Copel JA. Point-of-care ultrasonography. N Engl J Med. 2011 Feb 24;364(8):749-57. doi: 10.1056/NEJMra0909487. No abstract available. PMID 21345104
- [Background] Dietrich CF, Goudie A, Chiorean L, Cui XW, Gilja OH, Dong Y, Abramowicz JS, Vinayak S, Westerway SC, Nolsoe CP, Chou YH, Blaivas M. Point of Care Ultrasound: A WFUMB Position Paper. Ultrasound Med Biol. 2017 Jan;43(1):49-58. doi: 10.1016/j.ultrasmedbio.2016.06.021. Epub 2016 Jul 26. PMID 27472989
- [Background] Wagner M, Shen-Wagner J, Zhang KX, Flynn T, Bergman K. Point-of-Care Ultrasound Applications in the Outpatient Clinic. South Med J. 2018 Jul;111(7):404-410. doi: 10.14423/SMJ.0000000000000835. PMID 29978225
- [Background] Échographie ciblée pour les cliniciens de soins de première ligne [Internet]. Département de médecine de famille. [Internet]. [cité 1 mai 2020]. Disponible sur: https://www.mcgill.ca/familymed/fr/formation/programme-residence/echographie-ciblee-pour-les-cliniciens-de-soins-de-premiere-ligne
- [Background] Bécotte G, Garner M, Lanctôt J-F, Parent MC. Position conjointe de l'Association des médecins d'urgence du Québec (AMUQ) et de l'Association des spécialistes en médecine d'urgence du Québec (ASMUQ) adoptée le 7 novembre 2012. :16.
- [Background] Mayordomo-Colunga J, Gonzalez-Cortes R, Bravo MC, Martinez-Mas R, Vazquez-Martinez JL, Renter-Valdovinos L, Conlon TW, Nishisaki A, Cabanas F, Bilbao-Sustacha JA, Oulego-Erroz I. [Point-of-care ultrasound: Is it time to include it in the paediatric specialist training program?]. An Pediatr (Engl Ed). 2019 Sep;91(3):206.e1-206.e13. doi: 10.1016/j.anpedi.2019.06.012. Epub 2019 Aug 6. Spanish. PMID 31395389
- [Background] Torres-Macho J, Aro T, Bruckner I, Cogliati C, Gilja OH, Gurghean A, Karlafti E, Krsek M, Monhart Z, Muller-Marbach A, Neves J, Sabio R, Serra C, Smallwood N, Tana C, Uyaroglu OA, Von Wowern F, Bosch FH; EFIM s ultrasound working group.. Point-of-care ultrasound in internal medicine: A position paper by the ultrasound working group of the European federation of internal medicine. Eur J Intern Med. 2020 Mar;73:67-71. doi: 10.1016/j.ejim.2019.11.016. Epub 2019 Dec 11. PMID 31836177
- [Background] Bhagra A, Tierney DM, Sekiguchi H, Soni NJ. Point-of-Care Ultrasonography for Primary Care Physicians and General Internists. Mayo Clin Proc. 2016 Dec;91(12):1811-1827. doi: 10.1016/j.mayocp.2016.08.023. Epub 2016 Nov 5. PMID 27825617
- [Background] Liu RB, Donroe JH, McNamara RL, Forman HP, Moore CL. The Practice and Implications of Finding Fluid During Point-of-Care Ultrasonography: A Review. JAMA Intern Med. 2017 Dec 1;177(12):1818-1825. doi: 10.1001/jamainternmed.2017.5048. PMID 29059269
- [Background] Vinayak S, Sande J, Nisenbaum H, Nolsoe CP. Training Midwives to Perform Basic Obstetric Point-of-Care Ultrasound in Rural Areas Using a Tablet Platform and Mobile Phone Transmission Technology-A WFUMB COE Project. Ultrasound Med Biol. 2017 Oct;43(10):2125-2132. doi: 10.1016/j.ultrasmedbio.2017.05.024. Epub 2017 Jul 14. PMID 28716434
- [Background] Ma IWY, Arishenkoff S, Wiseman J, Desy J, Ailon J, Martin L, Otremba M, Halman S, Willemot P, Blouw M; Canadian Internal Medicine Ultrasound (CIMUS) Group*. Internal Medicine Point-of-Care Ultrasound Curriculum: Consensus Recommendations from the Canadian Internal Medicine Ultrasound (CIMUS) Group. J Gen Intern Med. 2017 Sep;32(9):1052-1057. doi: 10.1007/s11606-017-4071-5. Epub 2017 May 11. PMID 28497416
- [Background] Kimura BJ. Point-of-care cardiac ultrasound techniques in the physical examination: better at the bedside. Heart. 2017 Jul;103(13):987-994. doi: 10.1136/heartjnl-2016-309915. Epub 2017 Mar 4. PMID 28259843
- [Background] Arora S, Cheung AC, Tarique U, Agarwal A, Firdouse M, Ailon J. First-year medical students use of ultrasound or physical examination to diagnose hepatomegaly and ascites: a randomized controlled trial. J Ultrasound. 2017 Aug 19;20(3):199-204. doi: 10.1007/s40477-017-0261-6. eCollection 2017 Sep. PMID 28900520
- [Background] Buonsenso D, Pata D, Chiaretti A. COVID-19 outbreak: less stethoscope, more ultrasound. Lancet Respir Med. 2020 May;8(5):e27. doi: 10.1016/S2213-2600(20)30120-X. Epub 2020 Mar 20. No abstract available. PMID 32203708
- [Background] Hocine S. Part de l'échoscopie dans la pratique de l'échographie par les médecins généralistes français. Faculté de sciences médicales et paramédicales de Marseille; 2019.
- [Background] Delannoy Q. Quel est l'impact diagnostique et thérapeutique de l'échoscopie en pratique courante de Médecine Générale : Étude observationnelle et transversale. [Thèse d'exercice]. Sorbonne Université; 2018.
- [Background] Sorensen B, Hunskaar S. Point-of-care ultrasound in primary care: a systematic review of generalist performed point-of-care ultrasound in unselected populations. Ultrasound J. 2019 Nov 19;11(1):31. doi: 10.1186/s13089-019-0145-4. PMID 31749019
- [Background] Andersen CA, Davidsen AS, Brodersen J, Graumann O, Jensen MB. Danish general practitioners have found their own way of using point-of-care ultrasonography in primary care: a qualitative study. BMC Fam Pract. 2019 Jun 28;20(1):89. doi: 10.1186/s12875-019-0984-x. PMID 31253102
- [Background] Lokkegaard T, Todsen T, Nayahangan LJ, Andersen CA, Jensen MB, Konge L. Point-of-care ultrasound for general practitioners: a systematic needs assessment. Scand J Prim Health Care. 2020 Mar;38(1):3-11. doi: 10.1080/02813432.2020.1711572. Epub 2020 Jan 20. PMID 31955658
- [Background] Rempell JS, Saldana F, DiSalvo D, Kumar N, Stone MB, Chan W, Luz J, Noble VE, Liteplo A, Kimberly H, Kohler MJ. Pilot Point-of-Care Ultrasound Curriculum at Harvard Medical School: Early Experience. West J Emerg Med. 2016 Nov;17(6):734-740. doi: 10.5811/westjem.2016.8.31387. Epub 2016 Sep 12. PMID 27833681
- [Background] American Academy of Family Physicians. Recommended Curriculum Guidelines for Family Medicine Residents. Point of Care Ultrasound [Internet]. [cité 28 avr 2020]. Disponible sur: https://www.aafp.org/dam/AAFP/documents/medical_education_residency/program_directors/Reprint290D_POCUS.pdf
- [Background] Bornemann P. Assessment of a Novel Point-of-Care Ultrasound Curriculum's Effect on Competency Measures in Family Medicine Graduate Medical Education. J Ultrasound Med. 2017 Jun;36(6):1205-1211. doi: 10.7863/ultra.16.05002. Epub 2017 Feb 16. PMID 28206672
- [Background] Hoppmann RA, Rao VV, Bell F, Poston MB, Howe DB, Riffle S, Harris S, Riley R, McMahon C, Wilson LB, Blanck E, Richeson NA, Thomas LK, Hartman C, Neuffer FH, Keisler BD, Sims KM, Garber MD, Shuler CO, Blaivas M, Chillag SA, Wagner M, Barron K, Davis D, Wells JR, Kenney DJ, Hall JW, Bornemann PH, Schrift D, Hunt PS, Owens WB, Smith RS, Jackson AG, Hagon K, Wilson SP, Fowler SD, Catroppo JF, Rizvi AA, Powell CK, Cook T, Brown E, Navarro FA, Thornhill J, Burgis J, Jennings WR, McCallum JB, Nottingham JM, Kreiner J, Haddad R, Augustine JR, Pedigo NW, Catalana PV. The evolution of an integrated ultrasound curriculum (iUSC) for medical students: 9-year experience. Crit Ultrasound J. 2015 Dec;7(1):18. doi: 10.1186/s13089-015-0035-3. Epub 2015 Nov 21. PMID 26589313
- [Background] Andersen CA, Holden S, Vela J, Rathleff MS, Jensen MB. Point-of-Care Ultrasound in General Practice: A Systematic Review. Ann Fam Med. 2019 Jan;17(1):61-69. doi: 10.1370/afm.2330. PMID 30670398
- [Background] Steinmetz P, Oleskevich S. The benefits of doing ultrasound exams in your office. J Fam Pract. 2016 Aug;65(8):517-23. PMID 27660835
- [Background] Van Gansbeke V. [Sonography : a future imaging modality for the general practitioner ?]. Rev Med Brux. 2018;37(4):205-213. French. PMID 30320979
- [Background] Bornemann P, Jayasekera N, Bergman K, Ramos M, Gerhart J. Point-of-care ultrasound: Coming soon to primary care? J Fam Pract. 2018 Feb;67(2):70-80. PMID 29400896
- [Background] Myklestul HC, Skonnord T, Brekke M. Point-of-care ultrasound (POCUS) in Norwegian general practice. Scand J Prim Health Care. 2020 Jun;38(2):219-225. doi: 10.1080/02813432.2020.1753385. Epub 2020 Apr 21. PMID 32314640
- [Background] Zayyan M. Objective structured clinical examination: the assessment of choice. Oman Med J. 2011 Jul;26(4):219-22. doi: 10.5001/omj.2011.55. PMID 22043423
- [Background] Todsen T, Tolsgaard MG, Olsen BH, Henriksen BM, Hillingso JG, Konge L, Jensen ML, Ringsted C. Reliable and valid assessment of point-of-care ultrasonography. Ann Surg. 2015 Feb;261(2):309-15. doi: 10.1097/SLA.0000000000000552. PMID 24509198
- [Background] Wild D, Grove A, Martin M, Eremenco S, McElroy S, Verjee-Lorenz A, Erikson P; ISPOR Task Force for Translation and Cultural Adaptation. Principles of Good Practice for the Translation and Cultural Adaptation Process for Patient-Reported Outcomes (PRO) Measures: report of the ISPOR Task Force for Translation and Cultural Adaptation. Value Health. 2005 Mar-Apr;8(2):94-104. doi: 10.1111/j.1524-4733.2005.04054.x. PMID 15804318
- [Background] Lemanissier M. L'échographe, deuxième stéthoscope du médecin généraliste ? Validation d'une première liste d'indications d'échographies réalisables par le médecin généraliste. [Thèse d'exercice]. Université Paul Sabatier Toulouse III; 2013.
- [Background] Aakjaer Andersen C, Brodersen J, Davidsen AS, Graumann O, Jensen MBB. Use and impact of point-of-care ultrasonography in general practice: a prospective observational study. BMJ Open. 2020 Sep 17;10(9):e037664. doi: 10.1136/bmjopen-2020-037664. PMID 32948563

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: GPs were recruited as investigators. Investigators had to include patients undergoing POCUS in the study.
Groups:
- Patients With Physical Examination Before and After Ultrasound: Patients were recruited by GPs (investigators) There was no intervention in this group.
Period: Overall Study
Arm/Group | Patients With Physical Examination Before and After Ultrasound
Started | 655
Completed | 655
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Physical Examination With Ultrasound: This group included patients that were examined by GPs and had a point-of-care ultrasound (POCUS) during the consultation. There was no intervention in this group. The GPs used POCUS during their consultations as routine practice.
Arm/Group | Physical Examination With Ultrasound
Number analyzed (Participants) | 655
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 46 [32 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 412
  Male | 243
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Change in the Diagnosis After POCUS Examination
Description: GPs will register their diagnoses before and after the use of POCUS and a change in diagnosis will be described
  * one main diagnostic hypothesis
  * other diagnostic hypotheses After the use of POCUS, the GPs are asked if these diagnoses have changed and specify.
Time Frame: 20 to 30 minute consultation
Population: In the final analytic cohort of 655 patients, a time-log of more than 60 sec before and after POCUS was registered for 577 patients.
Measure: Count of Participants; unit: Participants
Groups:
- Physical Examination of Patients With Ultrasound: This group included patients that were examined by GPs and had a point-of-care ultrasound (POCUS) during the consultation. There was no intervention in this group. The GPs used POCUS during their consultations as routine practice.
  Patients with a time-log of more than 60 sec before and after POCUS were included in the before-after comparison.
Arm/Group | Physical Examination of Patients With Ultrasound
Number analyzed (Participants) | 577
Participants | 397

2. Primary Outcome: Number of Patients With Change in Diagnostic Confidence
Description: The GPs are asked to register any change in their confidence in the diagnostic hypothesis after the use of POCUS by choosing one of the following variables on an ordinal scale: increased confidence, more confident, unchanged confidence, less confident, reduced confidence
Time Frame: 30 minutes
Population: In the final cohort of 655 patients a time-log of more than 60 sec before and after POCUS was registered for 577 patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Physical Examination of Patients With Ultrasound
Number analyzed (Participants) | 577
Participants | 552

3. Primary Outcome: Number of Patients With Change in the Referral Plan
Description: Before using POC-US:
  * acute admission to hospital
  * subacute referral to hospital
  * normal referral to hospital
  * subacute referral to specialist
  * normal referral to specialist
  * referral for radiology
  * other referral (e.g. to physiotherapist, etc)
  * follow-up in the clinic
  * no plan for follow-up
  * other After using POC-US the GP is shown the "before POC-US plan for the patient" and asked if this plan has changed. If the plan has changed, the GP is asked to specify.
Time Frame: 20 to 30 minute consultation
Measure: Count of Participants; unit: Participants
Arm/Group | Physical Examination of Patients With Ultrasound
Number analyzed (Participants) | 577
Participants | 363

4. Primary Outcome: Number of Patients With Change in the Planned Treatment
Description: The GPs register their planned treatment before POCUS by choosing one or more of the following categorical variables:
  * medical treatment
  * non-medical treatment
  * no treatment
  * other After using POCUS, the GP is shown the "before POC-US planned treatment for the patient" and asked if this planned treatment has changed. If the planned treatment has changed, the GP is asked to specify.
Time Frame: 20 to 30 minute consultation
Measure: Count of Participants; unit: Participants
Arm/Group | Physical Examination of Patients With Ultrasound
Number analyzed (Participants) | 577
Participants | 215

ADVERSE EVENTS:
Time Frame: 0 min, adverse events were not collected
Description: There was no intervention in this study, therefore there was no assessment of adverse effects for patients included in the study during their consultation of 20-30 minutes.
Groups:
- Patient Physical Examination With Ultrasound: This group included patients that were examined by GPs and had a point-of-care ultrasound (POCUS) during the consultation. There was no intervention in this group. The GPs used POCUS during their consultations as routine practice.
Arm/Group | Patient Physical Examination With Ultrasound
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2025-05-22): https://cdn.clinicaltrials.gov/large-docs/70/NCT04583670/Prot_000.pdf
  • Statistical Analysis Plan (2025-05-22): https://cdn.clinicaltrials.gov/large-docs/70/NCT04583670/SAP_001.pdf